CLINICAL TRIAL: NCT05185791
Title: Feasibility and Clinical Results of Implementation of ERAS® Guidelines for Cytoreductive Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy: an International Prospective Cohort Study
Brief Title: ERAS® Guidelines Validation of CRS With or Without HIPEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 436
Record Dates: First submitted 2021-11-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Peritoneal Diseases
Keywords: CRS; HIPEC; ERAS®; Guidelines; Peritoneal metastasis; Colorectal; Gastric; ovarian; Peritoneal mesothelioma; Pseudomyxoma peritonei
MeSH Terms: conditions — Peritoneal Diseases; Pseudomyxoma Peritonei

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-ERAS® implementation phase: * Current clinical practice
  * Current perioperative management
  * All consecutive patients included for CRS+-HIPEC treatment
  * Period of inclusion : 3 months (01.10.2021 - 31.12.2021)
  * Survey of intended changes in clinical practice will be sent to each leader center
  No specific intervention. Only descriptive recordings of pre-intra-post-operative clinical endpoints ("ERAS® core items") and demographic parameters.
  Clinical and surgical outcomes will be recorded until 30 postoperative days (POD). Functional recovery parameters will be recorded for the first 5 POD
  Interventions: Other: Pre-ERAS® phase (current clinical practice)
- Post-ERAS® implementation phase: * After implementation 2 months of delay before starting the recordings
  * Clinical practice and perioperative management with new practice according guidelines and local commitment for the new change
  * All consecutive patients included for CRS±HIPEC treatment
  * Period of inclusion : 3 months (01.03.2022 - 31.05.2022)
  * Max 2 months of delay allowed between the two phases
  Intervention will take place during an implementation period of 2 months. This period will let the centers to set the newly implemented clinical practices.
  After that, the remaining 3 months of the study will consist in descriptive recordings of pre-intra and post-operative clinical endpoints and demographic parameters ("ERAS® core items").
  Clinical and surgical outcomes will be recorded until 30 postoperative days (POD). Functional recovery parameters will be recorded for the first 5 POD.
  Interventions: Other: Post-ERAS® implementation phase

INTERVENTIONS:
Other: Pre-ERAS® phase (current clinical practice) — Descriptive recordings of pre-intra-post-operative clinical endpoints and demographic parameters.
  Groups: Pre-ERAS® implementation phase
Other: Post-ERAS® implementation phase — Descriptive recordings of pre-intra-post-operative clinical endpoints and demographic parameters.
  Groups: Post-ERAS® implementation phase

SUMMARY:
Enhanced recovery after surgery (ERAS®) pathways have been shown to considerably reduce complications, length of stay and costs after most of surgical procedures by standardised application of best evidence-based perioperative care. Recently an international panel of expert have succeeded to elaborate dedicated recommendations for cytoreductive surgery (CRS) ± hyperthermic intraperitoneal chemotherapy (HIPEC) in a two-part series of guidelines based on expert consensus (Hübner et al., EJSO, 2020). The aim of this prospective validation study was therefore to study acceptance, feasibility and clinical results of these guidelines in clinical practice.

Hypothesis of the study: Introduction of ERAS® guidelines is feasible and safe. Increasing compliance with ERAS® guidelines (after implementation) will improve recovery and early clinical outcomes of patients undergoing CRS/HIPEC.

DETAILED DESCRIPTION:
The study includes two succesive phases interrupted by a stage to implement ERAS® guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults female and male patients (> 18 year-old)
* Peritoneal cancer from colorectal, ovarian, gastric, appendix origin and primitive peritoneal cancer (peritoneal mesothelioma)
* Multidisciplinary team meeting validation for CRS/HIPEC
* Informed and signed surgical consent

Exclusion Criteria:

* Patients without peritoneal cancer
* Patients with peritoneal cancer and extended extraperitoneal metastases contraindicating for CRS with or without HIPEC
* No informed consent signed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults patients suffering from cancer with peritoneal cancer eligible for surgery after passing a multidisciplinary team validation requiring CRS with or without HIPEC.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Compliance of ERAS® guidelines | 3 months
  Post-ERAS® implementation phase: compliance rate towards the relevant core items from ERAS guidelines

SECONDARY OUTCOMES:
Acceptance and feasibility of ERAS® guidelines | 3 months
  Pre-ERAS® phase (current clinical practice): current compliance rate towards the ERAS guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Glehen, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States
- University of Calgary, Arnie Charbonneau Cancer Institute, Calgary, Alberta, Canada
- Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hubner M, Kusamura S, Villeneuve L, Al-Niaimi A, Alyami M, Balonov K, Bell J, Bristow R, Guiral DC, Fagotti A, Falcao LFR, Glehen O, Lambert L, Mack L, Muenster T, Piso P, Pocard M, Rau B, Sgarbura O, Somashekhar SP, Wadhwa A, Altman A, Fawcett W, Veerapong J, Nelson G. Guidelines for Perioperative Care in Cytoreductive Surgery (CRS) with or without hyperthermic IntraPEritoneal chemotherapy (HIPEC): Enhanced recovery after surgery (ERAS(R)) Society Recommendations - Part I: Preoperative and intraoperative management. Eur J Surg Oncol. 2020 Dec;46(12):2292-2310. doi: 10.1016/j.ejso.2020.07.041. Epub 2020 Aug 25. PMID 32873454
- [Result] Hubner M, Kusamura S, Villeneuve L, Al-Niaimi A, Alyami M, Balonov K, Bell J, Bristow R, Guiral DC, Fagotti A, Falcao LFR, Glehen O, Lambert L, Mack L, Muenster T, Piso P, Pocard M, Rau B, Sgarbura O, Somashekhar SP, Wadhwa A, Altman A, Fawcett W, Veerapong J, Nelson G. Guidelines for Perioperative Care in Cytoreductive Surgery (CRS) with or without hyperthermic IntraPEritoneal chemotherapy (HIPEC): Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations - Part II: Postoperative management and special considerations. Eur J Surg Oncol. 2020 Dec;46(12):2311-2323. doi: 10.1016/j.ejso.2020.08.006. Epub 2020 Aug 13. PMID 32826114